CLINICAL TRIAL: NCT02930499
Title: A Prospective, Randomized, Controlled, Longitudinal Study Using Repeated Measures Design to Evaluate a Hyaluronic Acid Extracellular Matrix (Hyalomatrix®) in the Management of Chronic Venous Ulcers
Brief Title: Effect of Hyaluronic Acid ECM on Venous Ulcers
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator relocation
Sponsor: Calvary Hospital, Bronx, NY (Other)
Responsible Party: Principal Investigator, Oscar M. Alvarez, PhD, Director Wound Care Center, Calvary Hospital, Bronx, NY
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML-HM-0115-VLU
Record Dates: First submitted 2016-09-01; First posted 2016-10-12 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Venous Ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic Acid ECM (Hyalomatrix) (Experimental): Hyalomatrix ECM will be applied to the target ulcer once weekly
  Interventions: Device: Hyalomatrix extra-cellular matrix
- Non-Adherent wound dressing (Mepilex) (Active Comparator): Mepilex wound dressing will be applied to the target ulcer once weekly
  Interventions: Device: Mepilex wound dressing

INTERVENTIONS:
Device: Hyalomatrix extra-cellular matrix — An exta-cellular matrix made from hyaluronic acid
  Arms: Hyaluronic Acid ECM (Hyalomatrix)
Device: Mepilex wound dressing — A siliconized non-adhesive foam wound dressing
  Other Names: non-adhesive foam wound dressing
  Arms: Non-Adherent wound dressing (Mepilex)

SUMMARY:
The purpose of this pilot study is to compare the incidence and rate of wound healing in subjects with venous ulcers treated with an extracellular matrix composed of hyaluronic acid plus compression therapy as compared to standard care. The study also intends to follow the subjects for a 16-week period in order to evaluate ulcer recurrence within treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18-85 years of age with chronic venous insufficiency (CVI) and the presence of venous ulceration for longer than 2 months
2. Subject and/or caregiver must be willing and able to tolerate multi-layered compression bandages
3. Study subject must be reliable, responsible and able to visit the clinic weekly for the full 16 week period.

Exclusion Criteria:

1. Ulcers of non-venous etiology
2. Subject has a known sensitivity to hyaluronic acid
3. Presence of wound infection as determined by clinical signs and symptoms
4. Subject has any evidence of peripheral arterial disease (PAD)
5. Subject has received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within two weeks of screening date.
6. Pregnancy or lactation at time of treatment.
7. Subject is currently receiving or has received radiation or chemotherapy within 3 months of randomization.
8. Subject currently enrolled or participated within 30 days of baseline in another investigational device, drug or biological trial.
9. History of alcohol or drug abuse.
10. Subject allergic to a broad spectrum of primary & secondary dressing materials, including occlusive dressings and the adhesives on such dressings.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Effect of Hyalomatrix® plus standard care on the incidence of wound healing | 16 weeks

SECONDARY OUTCOMES:
Rate of wound healing by decrease in ulcer surface area Incidence of 50% wound healing by 4 weeks Reduced VLU recurrence after healing | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Alvarez, PhD, Principal Investigator — Program Director, Vascular and Wound Care Center, University Hospital, Newark, NJ
Locations (1):
- Vascular and Wound Care Center, University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided